CLINICAL TRIAL: NCT06265142
Title: Clean Catch Urine Feasibility and Contamination Rate Compared to Bladder Catheterization Urine in Pre-Continent Children: Randomized Control Trial
Brief Title: Clean Catch Urine Feasibility and Contamination Rate Compared to Bladder Catheterization Urine in Pre-Continent Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Sulayyem Saleh Al Harsousi, Principal Investigator, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MoH/CSR/23/26368
Record Dates: First submitted 2024-01-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Urinary Tract Infections
Keywords: clean catch urine; bladder massage; bladder catheterization; contamination rate
MeSH Terms: conditions — Urinary Tract Infections | interventions — Urinary Catheterization

STUDY DESIGN:
Intervention Model Description: Patient will be assessed in triage and cases to be included in the study as per the inclusion criteria, after that patients will be randomized using computerized block randomization technique into two groups. Then, patients will be assigned to a bed, pulse oximetry to be applied, data collection sheet to be filled, confirm that infant had good feeding/ didn't pass urine over last 20 minutes and proper cleaning to be done. The next step will be, collecting urine sample according to randomization group. Group A patients (control group), urine to be collected by standardized catheterization technique while group B by standard CCU technique. Meanwhile, time of each procedure to be documented. Regarding group B , after collecting urine by CCU , we recommend to collect another sample by catheterization to guide the management and antibiotic choice.
Who Masked: Outcomes Assessor
Masking Description: The statistician who will analyze the data will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheterization (Other): Group A: is the control group, participant will undergo bladder catheterization. (The standard practice)
  Interventions: Procedure: Bladder catheterization
- Clean Catch (Experimental): Group B: is the experimental group, participant will undergo clean catch urine via bladder massage technique.
  Interventions: Procedure: clean catch urine via bladder massage technique

INTERVENTIONS:
Procedure: Bladder catheterization — Participant will undergo the standard bladder catheterization for urine collection
  Arms: Catheterization
Procedure: clean catch urine via bladder massage technique — Participant will undergo clean catch urine via bladder massage technique
  Arms: Clean Catch

SUMMARY:
Introduction: Urinary tract infections (UTIs) are a common source of infection in children, accounting for a significant proportion of visits every year. Diagnosing UTIs requires obtaining a urine specimen, which can be collected using four methods: invasive techniques, such as suprapubic aspiration and urethral bladder catheterization, and noninvasive techniques, such as sterile bag and clean catch. However, catheterization can be a painful and invasive procedure, particularly in young infants who are less cooperative, and sometimes tends to be rejected by parents.

Given the availability of alternative methods with comparable contamination rates, we aim to investigate the feasibility and contamination rate of clean catch urine compared to bladder catheterization, as well as secondary outcomes such as pain scores, parental satisfaction, and time required to collect urine for each technique.

Methods: To achieve this, we will conduct a randomized control trial in precontinent pediatric patients. A pilot study with 40 samples in each arm will be conducted since there is no prior information about contamination rates in our setting. A well-designed and labeled data collection sheets will be used for data collection, and the data will be entered using EPI-data software. Statistical analysis will be performed using IBM SPSS statistics.

Aim: The main aim of this study is to introduce clean catch urine (bladder massage technique) to our setting, and to compare its feasibility with the bladder catheterization which is the standard practice.

Patient Population: young infants from 0 to 6 months of age

Intervention: There will be two groups:

1. Group A (Experimental group):Urine samples will be collected using the clean catch urine method (bladder massage technique).
2. Group B (Control group): Urine samples will be collected using the standard bladder catheterization method.

Clinical Measurement: All collected urine samples will be labeled and sent to the laboratory. All results will be retrieved from the medical records. Direct measurement will be for the duration of the procedures in both experiment and control group (stopwatch will be used). Pain score (Neonatal Infant Pain Scale) and parental satisfaction survey will be filled at the time of the procedure.

Outcome: Contamination rate and feasibility of both urine sampling techniques

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is a common source of infection in children. It accounts for 5 to 14 percent of visits by children every year. The overall prevalence is around 7% among different age subgroups of children. Several factors affect the prevalence of UTI including age, gender, and circumcision status.

The diagnosis of UTI requires obtaining a urine specimen from the patient. Generally, there are four methods used in collecting urine samples which can be categorized as invasive (such as suprapubic aspiration and urethral bladder catheterization) and noninvasive (such as Sterile bag and clean catch).

The selection of the urine collection technique is mainly determined by whether the patient is toilet-trained or not. In non-toilet-trained patients, urethral bladder catheterization or suprapubic aspiration can be used. The latter is having the least contamination rate in urine culture. Clean-catch urine is commonly used for toilet-trained patients. If the clinical assessment of febrile infants necessitates immediate antimicrobial therapy, urine culture should be obtained either by urethral bladder catheterization or suprapubic aspiration.

Previous observational studies showed approximately a 1 percent contamination rate using the suprapubic aspiration technique. In a prospective study done on premature infants it was found that the suprapubic aspiration technique resulted in increased pain and a higher probability of procedural failure compared to urethral bladder catheterization. According to American academy of pediatrics (AAP), for non-toilet trained children, it's advisable to gather a urine sample through methods like ureteral catheterization or suprapubic bladder aspiration, especially when a sample obtained using a perineal bag shows positive results on a dipstick test. The latest guideline from AAP recommends urine culture to be obtained via either SPA or bladder catheterization in pediatric patients aged between 8 to 60 days old, due to false positive results that can occur in the other urine collection techniques.

Urethral bladder catheterization carries a 6 to 12 percent of contamination rate. In regard clean catch urine method 16 to 63 percent of the contamination rate.

As outlined in the guideline in National Institute for Health and Care Excellence (NICE) guideline, to use clean catch urine wherever possible in pediatric patients below 16 years old. And to reserve bladder catheterization and suprapubic aspiration when noninvasive methods are not possible or practical.

previous literature demonstrated a safe and noninvasive technique to collect midstream clean-catch urine in infants. It was based on bladder stimulation and paravertebral lumbar massage. This technique yielded accurate and low contamination rates for infants below 90 days old. Moreover, the success rate was 86.3 percent, while the contamination rate was 5 percent. The safety and efficacy of the same stimulation technique in a neonatal intensive care unit setting were described in the literature. The median time to collect urine was 64 seconds. The success rate is 90 percent. However, some literature showed a lower success rate reaching 61 percent, possibly due to patients with a low oral intake that were not excluded from the study.

In the effort to reduce bladder catheterization in children, different techniques were introduced in the previous literature to improve the clean catch urine success rate as well as the contamination rate. Bladder and lumbar paravertebral massage maneuvers are a safe, time-saving technique that needs to be studied further.

In our setting, the recommendations from international guidelines are being followed. For non-toilet trained children suspected to have UTI, initial urine specimen for urine dipstick is collected by sterile bag or bladder catheterization. If the result of the urine dipstick came positive, then urine culture is obtained via bladder catheterization, if the initial specimen collected by the sterile bag. In addition, we lack the statistics of urine culture contamination in our laboratories.

The main aim of this study is to introduce clean catch urine (bladder massage technique) to our setting, and to compare its feasibility with the bladder catheterization which is the standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable infants.
* Require urine collection as part of their work-up in the emergency department.
* Age 0 to 6 months.

Exclusion Criteria:

* Parental refusal.
* Unstable hemodynamically young infants.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Urine culture contamination rate | After urine culture report (usually 2-3 days after urine collection)
  Urine culture contamination rate will be evaluated in both techniques used in the study which includes dividing the total number of contaminated urine culture sets by the total number of urine culture.
Parental satisfaction questionnaire | After the procedure immediately
  Parental satisfaction with the procedure techniques (in both arms) will be evaluated by a questionnaire.

SECONDARY OUTCOMES:
duration of the procedure | during each procedure
  duration of the procedure in both arms (in seconds)
Pain score | after the procedure immediately
  Pain score will be assessed by using Neonatal Infant Pain Scale (NIPS), values can range from 0 to 7. NIPS score interpretation 0-1: no pain; 2: mild pain; 3-4: moderate pain; 5-7: severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Lubna M Al Lawati, MD, Study Director — Oman Medical Speciality Board

IPD SHARING:
Plan to Share IPD: Undecided
Still undecided, as it is a pilot study. in the next main study, the IPD will be available.

REFERENCES:
- [Background] Shaikh N, Morone NE, Bost JE, Farrell MH. Prevalence of urinary tract infection in childhood: a meta-analysis. Pediatr Infect Dis J. 2008 Apr;27(4):302-8. doi: 10.1097/INF.0b013e31815e4122. PMID 18316994
- [Background] Nader, S. and Alejandro, H., 2021. Urinary tract infections in children: Epidemiology and risk factors. UpToDate, Waltham, MA, pp.1-19. (Accessed on January 01, 2023).
- [Background] Subcommittee on Urinary Tract Infection, Steering Committee on Quality Improvement and Management; Roberts KB. Urinary tract infection: clinical practice guideline for the diagnosis and management of the initial UTI in febrile infants and children 2 to 24 months. Pediatrics. 2011 Sep;128(3):595-610. doi: 10.1542/peds.2011-1330. Epub 2011 Aug 28. PMID 21873693
- [Background] Schroeder AR, Newman TB, Wasserman RC, Finch SA, Pantell RH. Choice of urine collection methods for the diagnosis of urinary tract infection in young, febrile infants. Arch Pediatr Adolesc Med. 2005 Oct;159(10):915-22. doi: 10.1001/archpedi.159.10.915. PMID 16203935
- [Background] Tosif S, Baker A, Oakley E, Donath S, Babl FE. Contamination rates of different urine collection methods for the diagnosis of urinary tract infections in young children: an observational cohort study. J Paediatr Child Health. 2012 Aug;48(8):659-64. doi: 10.1111/j.1440-1754.2012.02449.x. Epub 2012 Apr 27. PMID 22537082
- [Background] Labrosse M, Levy A, Autmizguine J, Gravel J. Evaluation of a New Strategy for Clean-Catch Urine in Infants. Pediatrics. 2016 Sep;138(3):e20160573. doi: 10.1542/peds.2016-0573. Epub 2016 Aug 19. PMID 27542848
- [Background] Al-Orifi F, McGillivray D, Tange S, Kramer MS. Urine culture from bag specimens in young children: are the risks too high? J Pediatr. 2000 Aug;137(2):221-6. doi: 10.1067/mpd.2000.107466. PMID 10931415
- [Background] Bogie AL, Sparkman A, Anderson M, Crittenden-Byers C, Barron M. Is There a Difference in the Contamination Rates of Urine Samples Obtained by Bladder Catheterization and Clean-Catch Collection in Preschool Children? Pediatr Emerg Care. 2021 Dec 1;37(12):e788-e790. doi: 10.1097/PEC.0000000000002578. PMID 34772880
- [Background] Ballouhey Q, Fourcade L, Couve-Deacon E, Cros J, Lescure V, Bahans C, Chainier D, Garnier F, Guigonis V. Urine Contamination in Nontoilet-trained and Uncircumcised Boys. Urology. 2016 Sep;95:171-4. doi: 10.1016/j.urology.2016.05.056. Epub 2016 Jun 8. PMID 27289027
- [Background] Badiee Z, Sadeghnia A, Zarean N. Suprapubic Bladder Aspiration or Urethral Catheterization: Which is More Painful in Uncircumcised Male Newborns? Int J Prev Med. 2014 Sep;5(9):1125-30. PMID 25317295
- [Background] Mattoo TK, Shaikh N, Nelson CP. Contemporary Management of Urinary Tract Infection in Children. Pediatrics. 2021 Feb;147(2):e2020012138. doi: 10.1542/peds.2020-012138. PMID 33479164
- [Background] Pantell RH, Roberts KB, Adams WG, Dreyer BP, Kuppermann N, O'Leary ST, Okechukwu K, Woods CR Jr; SUBCOMMITTEE ON FEBRILE INFANTS. Evaluation and Management of Well-Appearing Febrile Infants 8 to 60 Days Old. Pediatrics. 2021 Aug;148(2):e2021052228. doi: 10.1542/peds.2021-052228. Epub 2021 Jul 19. PMID 34281996
- [Background] National Institute for Health and Care Excellence. (2007). Urinary tract infection in under 16s: diagnosis and management. Clinical guideline.. nice. org. uk/guidance/cg54.
- [Background] Altuntas N, Tayfur AC, Kocak M, Razi HC, Akkurt S. Midstream clean-catch urine collection in newborns: a randomized controlled study. Eur J Pediatr. 2015 May;174(5):577-82. doi: 10.1007/s00431-014-2434-z. Epub 2014 Oct 17. PMID 25319844
- [Background] Herreros ML, Tagarro A, Garcia-Pose A, Sanchez A, Canete A, Gili P. Accuracy of a new clean-catch technique for diagnosis of urinary tract infection in infants younger than 90 days of age. Paediatr Child Health. 2015 Aug-Sep;20(6):e30-2. PMID 26435675
- [Background] Mulcrone AE, Parikh M, Ahmad FA. Reducing infant catheterization in the emergency department through clean-catch urine collection. J Am Coll Emerg Physicians Open. 2020 Aug 17;1(6):1533-1541. doi: 10.1002/emp2.12211. eCollection 2020 Dec. PMID 33392562

DOCUMENTS (2):
  • Study Protocol (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT06265142/Prot_000.pdf
  • Informed Consent Form (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT06265142/ICF_001.pdf